CLINICAL TRIAL: NCT01831934
Title: Metabolic and Immune Responses to TIV in Patients With Mitochondrial Disease
Brief Title: Responses to Influenza Vaccine in Patients With Mitochondrial Disorders (MELAS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cornelia L. Dekker, Professor, Pediatrics, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-18615; R21HD061709-01A1 (NIH)
Record Dates: First submitted 2013-03-19; First posted 2013-04-15 (Estimated); Results first posted 2017-04-21 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: MELAS Syndrome
Keywords: Mitochondrial disorder; Trivalent inactivated influenza vaccine; Adolescents and adults; Immune response; Metabolic response
MeSH Terms: conditions — MELAS Syndrome; Mitochondrial Diseases | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MELAS group:13-60 years of age. (Experimental): Fluzone® 2010-2011 Formula or 2011-2012 depending on year
  Interventions: Biological: Fluzone®
- Control Group: 18-65 years of age (Experimental): Fluzone® 2010-2011 Formula or 2011-2012 depending on year
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: Fluzone® — This vaccine is given intramuscularly, either the 2010-2011 or 2011-2012 vaccination was given as appropriate
  Other Names: trivalent inactivated influenza vaccine (TIV); FDA-licensed seasonal influenza vaccine

SUMMARY:
This pilot clinical study evaluated the safety and metabolic responses to a licensed inactivated seasonal influenza vaccine (TIV) in mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes syndrome (MELAS) volunteers and controls.

DETAILED DESCRIPTION:
This pilot clinical study evaluated the safety and metabolic responses to a licensed inactivated seasonal influenza vaccine (TIV). This study will consist of two cohorts: MELAS syndrome volunteers (a specific identified disorder of mitochondrial dysfunction: mitochondrial encephalopathy, lactic acidosis, and stroke-like episodes) between 13-60 years OR adult control volunteers between 18-65 years of age. Both cohorts will receive the same treatment: a single vaccination with an FDA-licensed intramuscular seasonal trivalent inactivated influenza vaccine (TIV).

All participants will receive a single administration of a licensed influenza vaccine. Prior to vaccination, participants will provide information regarding health history and responses to health questionnaires. A blood sample and urine specimen were collected prior to vaccination, and at 6 hours, 5-7 days and 26-30 days post-immunization.

ELIGIBILITY:
Inclusion Criteria:Inclusion criteria include:

* Age between 13-60 years for MELAS volunteers OR age between 18-65 years for adult control volunteers. Control volunteers will be age-matched +/-5 years to enrolled MELAS volunteers. If the MELAS volunteer has diabetes and uses insulin daily, their control will be an adult with diabetes who uses insulin daily.
* General good health at time of enrollment
* Willing and able to sign Informed Consent
* Available for follow-up for the planned duration of the study
* Acceptable medical history by screening evaluation and brief clinical assessment
* All female participants of childbearing potential must use an acceptable method of contraception and not become pregnant for the duration of the clinical phase of the study (approximately 1 month to completion of Visit 4). (Acceptable contraception may include but is not limited to implants, injectables, combined oral contraceptives, effective intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner).

Exclusion Criteria:Exclusion criteria will include:

* Allergy to egg or egg products or allergy to vaccine components, including thimerosal
* Active systemic or serious concurrent illness, including febrile illness, within the 3 days prior to study vaccination
* History of immunodeficiency, known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* Blood pressure >150 systolic or >95 diastolic at Visit 1.
* Hospitalization in the past year for congestive heart failure or emphysema.
* History of chronic Hepatitis B or C.
* Recent or current use of immunosuppressive medication, including glucocorticoids (corticosteroid nasal sprays are permissible).
* Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
* Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Receipt of blood or blood products within the past 6 months
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* Inactivated vaccine 14 days prior to vaccination or live, attenuated vaccine within 60 days of vaccination
* History of Guillain-Barré Syndrome
* Pregnant or lactating woman
* Use of investigational agents within 30 days prior to enrollment
* Donation of the equivalent of a unit of blood within 6 weeks prior to enrollment
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2010-09; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Gregory M Enns, MBChB, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MELAS Group:13-60 Years of Age.; Control Group: 18-65 Years of Age: Fluzone® 2011-2012 Formula
  Fluzone® 2011-2012 Formula: Quadrivalent inactivated influenza vaccine given given intramuscularly in 0.5ml doses.
Period: Overall Study
Arm/Group | MELAS Group:13-60 Years of Age. | Control Group: 18-65 Years of Age
Started | 12 | 10
Completed | 11 (Volunteer consented but not enrolled after reporting a prior bad reaction to influenza vaccine.) | 10
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MELAS Group; Control Group: Fluzone®
  Fluzone®
- Total: Total of all reporting groups
Arm/Group | MELAS Group | Control Group | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.74 (8.06) | 37.39 (10.04) | 38.13 (8.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 9 | 20
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 4 | 13
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Clinical Safety of TIV Vaccine
Description: We will measure solicited local and systemic adverse events and SAEs for 1 month following immunization
Time Frame: Day 0 to Day28
Measure: Count of Participants; unit: Participants
Groups:
- MELAS Group; Control Group: Fluzone® 2011-2012 Formula
  Fluzone® 2011-2012 Formula: This vaccine is given intramuscularly
Arm/Group | MELAS Group | Control Group
Number analyzed (Participants) | 12 | 10
Participants
  Number of Adverse Events | 4 | 0
  Number of Severe Adverse Events | 0 | 0
  Number with no Adverse Events | 8 | 10

2. Other Pre Specified Outcome: Measurement of Intracellular Glutathione by Hi-D FACS (CD4 and CD8 T Cells) and Tandem Mass Spectrometry (Whole Blood)
Description: This method relies on the ability of intracellular glutathione S-transferases to tag GSH to bimane to yield a bimane-GS conjugate that fluoresces at 440 nm.
Time Frame: Day 0-Day28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days post immunization
Arm/Group | MELAS Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 4/12 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MELAS Group (N=12) | Control Group (N=10)
Seizure (Nervous system disorders) | 1 (3) | 0 (0) — A volunteer experienced 3 seizures lasting approximately 10 minutes. These were of the same type as his baseline seizures, but different in length and frequency. He was seen by his regular neurologist who left his medications unchanged.
Nasal Discharge (General disorders) | 2 (2) | 0 (0)
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — report of occasional intermittent spasm of right jaw four days post vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No